CLINICAL TRIAL: NCT04029064
Title: Management of Prenatally Diagnosed Isolated Right Aortic Arch: the ARCADE Study
Brief Title: Management of Prenatally Diagnosed Isolated Right Aortic Arch
Acronym: ARCADE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Congeital heart disease explorations unit - UE3C Lowendal - Paris (Unknown); University Hospital, Rouen (Other); Nantes University Hospital (Other); University Hospital, Grenoble (Other); University Hospital, Bordeaux (Other); Clinique La louvère - Lille - France (Unknown); University Hospital, Tours (Other); University Hospital, Caen (Other); University Hospital, Toulouse (Other); Hospices Civils de Lyon (Other); University Hospital, Marseille (Other); Amiens University Hospital (Other); Martinique University Hospital (Unknown); Centre Hospitalier Universitaire Dijon (Other); Private cardiology practice, Massy (Unknown); Private cardiology practice, Marseille (Unknown); Private cardiology practice, Pontoise (Unknown); Private cardiology practice, Strasbourg (Unknown); Private cardiology practice, Brest (Unknown); Private cardiology practice, Rennes (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0146
Record Dates: First submitted 2019-04-25; First posted 2019-07-23 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-03

CONDITIONS: Isolated Right Aortic Arch
Keywords: right aortic arch; congenital heart disease; pediatrics; cardiology; prenatal diagnosis
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The existence of a right aortic arch integrates nosologically into the group of aortic vascular arch anomalies. In the majority of cases, a right aortic arch is associated with cono-truncal congenital heart diseases (CHD), such as tetralogy of Fallot, pulmonary atresia with ventricular septal defect, and truncus arteriosus. Sometimes, a right aortic arch can be isolated, with an incidence of 0.05% to 0.1 %. Therefore, an assessment of the anatomy is necessary because an isolated right aortic arch can be associated with an encircling aortic arch anomaly and may subsequently have a functional repercussion, creating a digestive obstacle (oesophageal compression) and/or a respiratory obstacle (tracheal compression).

Furthermore, indications for surgery in this type of abnormalities are not well-established.

The diagnosis of a vascular artery anomaly is currently mostly made prenatally, with increasing diagnostic accuracy. Indeed, the application of the "3VT view" (e.g. three vessels and tracheae view) in routine prenatal sonographic screening for CHD has contributed to a better identification of such anomalies.

Prenatal diagnosis of an isolated right aortic arch involves the identification of the following aspects: the existence of a left ductus arteriosus may relate to an increased risk of an encircling aortic arch anomaly at birth; the analysis of the different vessels of the aortic arch, which can be difficult because of the fetal circulation and the maternal-fetal conditions of the examination; and the absence of a thymus, which suggests the existence of a genetic anomaly, such as DiGeorge syndrome.

After birth, the evaluation of the functional repercussion of the anomaly remains complex. The incidence of secondary symptoms to encircling abnormalities is estimated at 25%, but varies according to the anomaly: it is very frequent in case of a double aortic arch, variable in case of a right aortic arch with left ductus arteriosus (from 9% to 47% in the literature), absent in case of right aortic arch with right ductus arteriosus. Postnatal echocardiography can only assess the existence of a right aortic arch and check ductus arteriosus closure. The complete anatomical diagnosis of a vascular artery anomaly can only be made by slice cardiac imaging (CT scan or MRI), but in practice these examinations are not routinely performed in the absence of neonatal symptoms.

The aim of this study is to evaluate the accuracy of prenatally diagnosed isolated right aortic arch in terms of anatomy and functional prognosis.

The secondary aims are :

* to specify the association of an isolated right aortic arch with a genetic anomaly,
* to define the role of CT scan in children prenatally diagnosed with right aortic arch, in terms of diagnosis, prognosis and follow-up,
* to evaluate the incidence of respiratory and digestive complications in the first year of life,
* to evaluate the indications for surgical management during the first year of life.

DETAILED DESCRIPTION:
Retrospective (from 2010 to 2019), multicentre, observational study carried out in the French national M3C network (complex CHD expert centers).

Patients with a prenatal diagnosis of isolated right aortic arch will be included. Patients with a right aortic arch associated with any CHD will be excluded, as well as patients whose parents refuse the use of medical data of their child.

The following data will be collected:

Clinical data:

* Functional signs of tracheal or esophageal compression in the first year of life.
* Association with a genetic syndrome.

Echocardiographic data:

* Prenatal: anatomical description of the aorta and supra-aortic trunks. Position of the ductus arteriosus, presence of a thymus.
* Postnatal: confirmation of the right aortic arch, absence of conotruncal CHD, closure of the ductus arteriosus.

If performing a chest CT scan in the first year of life:

* Reason: systematic or on symptoms,
* Age of realization,
* Anatomical analysis of the aortic arches,
* Concordance with antenatal diagnosis,
* Evaluation of the degree of tracheal compression,
* Screening for a vascular complication.

If performing an ante- or post-natal genetic sampling:

* Type of sampling if antenatal: amniocentesis or trophoblast biopsy,
* Type of analysis: karyotype, FISH, CGH array,
* Molecular diagnosis.

If performing a surgery during the first year of life:

* Indication: prophylactic or symptomatic,
* Type of intervention,
* Age at the intervention

ELIGIBILITY:
Inclusion criteria:

• Prenatal diagnosis of an isolated right aortic arch

Exclusion criteria:

* Association with any congenital heart disease according to the ACC-CHD (Orphanet) classification
* Postnatal diagnosis of an isolated right aortic arch
* Refusal of parents to use medical data

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with antenatal diagnosis of isolated right aortic arch
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between the antenatal description of isolated right aortic arch and the postnatal description and functional prognosis | 1 day
  Correlation between the antenatal description of isolated right aortic arch and the postnatal description and functional prognosis

SECONDARY OUTCOMES:
Rate of genetic anomaly with an isolated right aortic arch | 1 day
  Incidence of genetic anomaly with an isolated right aortic arch by specifying :
  * diagnosed retained
  * type of sampling : amniocentesis, trophoblast biopsy, blood test
  * type of analysis: karyotype, FISH, CGH array
Rate of realization of chest CT angiography before the first year of life with an isolated right aortic arch | 1 day
  If performing a chest CT scan the first year of life:
  * Reason: systematic or on symptoms
  * Age of realization
  * Anatomical analysis of the aortic arches
  * Concordance with antenatal diagnosis
  * Evaluation of the degree of tracheal compression
Rate of surgical repair during the first year of life after prenatal diagnosis of an isolated right aortic arch. | 1 day
  If performing a surgery the first year of life:
  * Indication: prophylactic or symptomatic
  * Type of intervention
  * Age at the intervention
Rate of respiratory and digestive complications in the first year of life. | 1 day
  Functional signs of tracheal or esophageal compression in the first year of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie GUILLAUMONT, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Guillaumont S, Vincenti M, Thomas F, Huguet H, Picot MC, Abassi H, Huby AC, Laux D, Thomas-Chabaneix J, Cohen L, Gavotto A, Amedro P; ARCADE study group. Implications of right aortic arch prenatal diagnosis: the multicentric nationwide ARCADE cohort. Arch Dis Child Fetal Neonatal Ed. 2025 Feb 21;110(2):138-144. doi: 10.1136/archdischild-2024-327242. PMID 38964845